CLINICAL TRIAL: NCT03306173
Title: COMET Study 1: Filter Ventilated Cigarette Substitution in the ETM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CigVent Proj-003; 1P01CA217806 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-10 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either use a ventilated or unventilated cigarette.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to either ventilated or unventilated cigarettes and will not be informed of their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilated cigarettes (Experimental): Participants in this ARM will be assigned to ~25% filter ventilation commercially available cigarettes.
  Interventions: Other: Commercially available cigarette
- Unventilated cigarettes (Experimental): Participants in this ARM will be assigned to ~0% filter ventilation commercially available cigarettes.
  Interventions: Other: Commercially available cigarette

INTERVENTIONS:
Other: Commercially available cigarette — Commercially available cigarette with either ~0% or ~25% filter ventilation. Menthol flavor will be available in both types.

SUMMARY:
Early attempts by the tobacco industry to develop "safer" cigarettes led to the widespread introduction of ventilation holes in cigarette filters; however, this design feature may instead increase smoking-related harm and make cigarettes more palatable. The overall goal of this project is to model regulatory restrictions banning cigarette filter ventilation and determine their effects on consumption of both cigarettes and a wide range of alternative tobacco products. Testing potential regulatory actions under controlled conditions will facilitate evidence-based policies that have a net benefit to health.

DETAILED DESCRIPTION:
Early attempts by the tobacco industry to develop "safer" cigarettes led to the widespread introduction of ventilation holes in cigarette filters; however, this design feature may instead increase smoking-related harm and make cigarettes more palatable. The overall goal of this project is to model regulatory restrictions banning cigarette filter ventilation and determine their effects on consumption of both cigarettes and a wide range of alternative tobacco products. Testing potential regulatory actions under controlled conditions will facilitate evidence-based policies that have a net benefit to health.

Detailed Description:

The duration of the experiment will be approximately 3 months. Participants will begin with an initial one week (approximately) exposure period to both unventilated and ventilated cigarettes as well as alternative nicotine products (e-cigarettes, snus, etc.) that will be made available throughout the experiment. Participants will be given the opportunity to sample both types of cigarettes and alternative nicotine products. In the following sessions, participants will alternate between Electronic Tobacco Marketplace (ETM) sessions and free exposure periods to their assigned cigarette, with weekly assessments throughout to track changes in smoking behavior and cigarette valuation. In total, participants will complete 10 experimental sessions (see Appendix B for experimental timeline figure). For the sake of clarity, session types are separated below. The consent and initial sessions may take place in the same or separate sessions.

At the beginning of the experiment, participants will be assigned to one of two groups: ventilated or unventilated. Group assignment will determine what cigarettes will be given to the participant after sessions in which they do not actually purchase their cigarettes of choice. Additionally, participants that typically smoke menthol cigarettes will be given a menthol version of their assigned cigarette. Cigarettes will be similar in design and will be labeled as Typa A or Type B.

At the initial session and throughout the study, urine samples may be collected and stored for testing (for tobacco use and pregnancy) and breath samples for carbon monoxide and alcohol. Self-report may be used in place of urine analyses on a case-by-case bases. Urine sample analyses for tobacco use may only take place at the VTCRI site.

Initial Assessment Session and Sampling (Session 1). First, participants will complete the consenting process. The first session will be an assessment session to collect information from participants on patterns and degree of tobacco and other substance use, perceptions of all cigarette types available in the ETM, as well as the results of behavioral and cognitive tasks that we think may inform or complement the results from the main study (see Appendix A for a complete list and descriptions).

Participants will also complete the initial sampling period following the initial sampling session. The goal of this period is to familiarize the participants with their randomly assigned cigarette as well as alternative nicotine products. After their assessment session, participants will be given a 7-day supply of ventilated and unventilated (3.5 days of venitlated and 3.5 days of unventialted) cigarettes and asked to use these cigarettes. The actual number of cigarettes delivered to each participant will be determined by multiplying their reported cigarettes smoked per day by 7. Therefore, the average minimum number of cigarettes that will be delivered is approximately 70 (10 cigarettes per day minimum to qualify to participate). They will be also be given a sample of the alternative nicotine products that will be made available during the Real-ETM sessions. Participants will be asked to report their favorite flavor of each product to sample. If the participant is naïve to the alternative nicotine product, they will be asked to estimate which product flavor they would prefer. To verify usage during this and all subsequent usage period (see below), participants will be asked to return spent cigarette filters in resealable bags we provide. However, while participants will be asked to smoke the cigarettes they are given and to not use any other cigarettes, they will only be asked to try the alternative nicotine products during the sampling period, they do not have to finish them. A subset of these spent filters will be randomly chosen and analyzed to permit correlation of mouth-level exposure to smoke constituents with differences in ETM purchasing behavior between ventilated and unventilated cigarettes. During this sampling period, participants will go about their daily lives, allowing them to sample these cigarettes in the social environment in which they typically operate. This "real-world" sampling period will serve to increase the generalizability of the results obtained in the ETM sessions. This duration of exposure was chosen to give participants time to begin to familiarize themselves with their assigned cigarettes. This will enable them to make informed purchasing decisions during the upcoming sessions.

Real Experimental Tobacco Marketplace Sessions (Sessions 2,6, and 10).

Following the initial sampling period, participants will complete a purchasing session in our realistic tobacco product marketplace. Participants will be seated in front of a computer to access an online marketplace with an interface similar to many online merchants. This will allow participants to browse through the products and add as many as they desire to the virtual shopping cart. Each product will have the price clearly displayed along with an image. Each ETM session will contain five pricing scenarios, in which we:

i. manipulate the price of participants' assigned cigarettes to assess demand in a context with no other products available; ii. manipulate the price of participants' non-assigned cigarettes to assess demand in a context with no other products available; iii. manipulate the price of both assigned and non-assigned cigarettes in unison to assess simple preference between the two; iv. manipulate the price of participants' assigned cigarettes while the price of non-assigned cigarettes remains constant to assess the degree to which assigned cigarettes substitute for non-assigned cigarettes;

a. In this task, alternative nicotine products (e.g., e-cigarettes, chew, etc.) may also be available for purchase at a constant price.

v. manipulate the price of participants' non-assigned cigarette while the price of assigned cigarettes remains constant to assess the degree to which non-assigned cigarettes substitute for assigned cigarettes.

a. In this task, alternative nicotine products (e.g., e-cigarettes, chew, etc.) may also be available for purchase at a constant price.

In each of these scenarios, the price-manipulated cigarettes will be available across a range of prices (e.g., $0.12, $0.25, $0.50, $1.00, $2.00, and $4.00). Price-constant cigarettes will be set to the median cigarette price in the community. Participants will use an experimentally provided income (proportional to their real-world tobacco consumption) to purchase from the ETM. At each price, participants will be asked to make seven days of tobacco-product purchases from the ETM. After all 5 scenarios are complete for their assigned cigarette, participants will receive the products they purchased from one randomly selected price. Participants will be well informed of these procedures prior to purchasing. For those seven days after marketplace sessions, participants will be asked to only use those products they have purchased from the tobacco marketplace, and to not purchase any outside tobacco products, to not sell or give away any of their purchases, and to not ask anybody else to purchase products for them. We will strongly encourage participants to follow these procedures, and to report any deviations from these procedures, which we will incorporate into our statistical analyses. If the participant does not spend their entire income, they will be allowed to keep the remainder. In this way, participants will be spending real money and incurring a financial cost for their purchases, leading to more realistic product selections. Following the seven days of using cigarettes obtained from the ETM, participants will again visit the lab to return any unused products and report the use of experimenter provided and non-experimenter provided tobacco products.

Extended Cigarette Exposure and Experimental Tobacco Marketplace Testing (Sessions 3, 4, 5, 7, 8, and 9).

Following the first session in the ETM and its associated period of tobacco product use, participants will begin periods of freely provided exposure to their assigned cigarette (ventilated or unventilated), alternating with two additional sessions in the ETM at regular intervals. The purpose of this additional exposure between discrete ETM assessments is so that we may examine the effects of sustained exposure to participants' assigned cigarettes at regular intervals. During the extended-exposure periods, participants will visit the lab every 7 days. At each of these sessions during extended-exposure periods, they will return any unused cigarettes, report the use of experimenter provided and non-experimenter provided tobacco products, receive cigarettes for the upcoming 7 days, and complete many of the assessments they completed at their initial assessment session.

Following sessions 5 and 9 (the sessions immediately before the Real ETM sessions) participants will be given 6 days of their assigned cigarettes and 1 day of the unassigned cigarettes in order to expose the participant to the unassigned cigarettes before the Real ETM session.

An abbreviated set of assessments will be collected on a weekly basis throughout the experiment (Appendix A) in addition to any additional scheduled session (e.g., Real ETM). These assessments will focus on measuring tobacco product use and measures of dependence and withdrawal, including a Timeline Follow-Back for the period since the last session, as well as product perceptions. We will also include a purely hypothetical version of the ETM (on non-real ETM sessions), in which participants do not receive products purchased to use outside the laboratory. Because these hypothetical ETM assessments can be repeated with greater frequency and without interrupting periods of continuous exposure to assigned cigarettes, data from hypothetical assessments will be used to inform determinations of the effects of time on valuation of ventilated and unventilated cigarettes in more detail than primary ETM assessments.

The study design focuses on comparing ventilated versus unventilated cigarette groups to determine the impact of cigarette filter ventilation on tobacco product selection, consumption, and potential substitution to alternative products.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker
* Stable mental and physical health
* Does not take medications that interfere with nicotine metabolism

Exclusion Criteria:

* Pregnant or lactating
* Immediate future plans to quit smoking

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, PHD, Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Results from research conducted under this project will be disseminated in several ways. Findings will be presented at national conferences for groups such as the Society for Research on Nicotine and Tobacco (SRNT) and the College on Problems of Drug Dependence (CPDD). Manuscripts will be written and submitted for publication in a timely manner in high-quality peer-reviewed journals, following the NIH Public Access Policy guidelines.
Time Frame: Data will be made available upon request after dissemination of results.
Access Criteria: Data requests will be reviewed by the principal investigator and data will be shared with the expectation of acknowledgment of funding source and primary study team.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants enrolled differs from those who started the study because, after providing informed consent, participants submitted a breath carbon monoxide (CO) sample to assess recent cigarette use. Participants were excluded from the study if their CO level was below 8 ppm, indicating no recent smoking. They consented and were assigned to an arm/group, however, they didn't begin the intervention they were assigned to.
Period: Overall Study
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Started | 68 | 68
Completed | 44 | 38
Not Completed | 24 | 30
Not completed — Lost to Follow-up | 16 | 23
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Discontinued | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes | Total
Number analyzed (Participants) | 44 | 38 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years of age] | 45.61 (11.21) | 43.16 (10.66) | 44.48 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 22 | 14 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 42 | 38 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 35 | 33 | 68
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 38 | 82
Cigarettes per day [Mean (Standard Deviation); unit: Number of cigarettes] — Number of cigarettes participants smoked per day
  Number of cigarettes | 19.91 (6.28) | 20.71 (7.38) | 20.28 (6.78)
PHR High Ventilated Cigarettes [Mean (Standard Deviation); unit: Scores on a scale] — The Perceived Health Risk (PHR) is a 10-point scale used to assess perceived disease risk, ranging from 1 (very low risk) to 10 (very high risk). Total scores range from 9 to 90 and higher scores reflect greater perceived health risk toward the disease. It is a 9-item scale. We summed all subscale scores for each participant, then summed all participants' scores and calculated the group's mean and standard deviation.
  Scores on a scale | 62.61 (22.44) | 49.00 (21.14) | 56.30 (22.76)
PHR Low Ventilated Cigarettes [Mean (Standard Deviation); unit: Scores on a scale] — The Perceived Health Risk (PHR) is a 10-point scale used to assess perceived disease risk, ranging from 1 (very low risk) to 10 (very high risk). Total scores range from 9 to 90 and higher scores reflect greater perceived health risk toward the disease. It is a 9-item scale. We summed all subscale scores for each participant, then summed all participants' scores and calculated the group's mean and standard deviation.
  Scores on a scale | 62.61 (22.99) | 49.76 (23.59) | 56.66 (24.01)
Fagerstrom Test for Cigarette Dependence [Mean (Standard Deviation); unit: Scores on a scale] — The Fagerstrom Test for Cigarette Dependence is a 6-item scale to assess cigarette dependence. Scores range from 0 to 10: 0 represents no dependence, 1-2 low dependence, 3-4 low to moderate dependence, 5-7 moderate dependence and 8-10 represents high dependence. We summed all participants scores and calculated the mean and standard deviation of the group.
  Scores on a scale | 3.93 (1.39) | 4.16 (1.42) | 4.04 (1.40)
QSU [Mean (Standard Deviation); unit: Scores on a scale] — The Questionnaire of Smoking Urges - Brief (QSU-Brief) is a 10-item measure used to assess craving to smoke. Participants rate each statement on a 7-point Likert scale, ranging from "strongly disagree" (1) to "strongly agree" (7). Total scores range from 10 to 70, with higher scores indicating a stronger urge to smoke. We summed each participant's responses to obtain total scores, then calculated the group mean and standard deviation.
  Scores on a scale | 43.98 (15.40) | 44.03 (14.10) | 44.00 (14.72)
RHQ [Mean (Standard Deviation); unit: Scores on a scale] — The Respiratory Health Questionnaire (RHQ) is a 4-item scale designed to assess respiratory issues. It uses a 10-point scale ranging from "None" to "Severe" to evaluate issues such as breathing difficulties, coughing, and lung irritation. Total scores range from 4 to 40 and higher scores represents poorer respiratory health. We summed all participants scores and calculated the mean and standard deviation of the group.
  Scores on a scale | 14.41 (7.08) | 12.05 (5.36) | 13.32 (6.42)
WISDM [Mean (Standard Deviation); unit: Scores on a scale] — The Wisconsin Inventory of Smoking Dependence Motives (WISDM) is a 68-item questionnaire with 13 subscales designed to assess various motives underlying smoking dependence. Respondents rate each item on a 7-point scale, ranging from 1 ("Not true of me at all") to 7 ("Extremely true of me"). The total scores range from 68 to 476 and higher scores represents higher tobacco dependence. We summed the subscales scores then we summed the resultant scores and calculated the mean and standard deviation of the group.
  Scores on a scale | 182.48 (51.95) | 180.53 (38.84) | 181.57 (46.07)
MNWS [Mean (Standard Deviation); unit: Scores on a scale] — The Minnesota Nicotine Withdrawal Scale (MNWS) is a self-report instrument designed to assess symptoms of nicotine withdrawal. Each item is rated on a 5-point scale ranging from 0 ("None") to 4 ("Severe"). Total scores range from 0 to 32 and higher scores represents severe withdrawal symptoms. We summed all participants scores and calculated the mean and standard deviation of the group.
  Scores on a scale | 15.25 (10.65) | 13.34 (8.87) | 14.37 (9.85)

OUTCOME MEASURES:

1. Primary Outcome: High Ventilated Cigarette Purchases
Description: Participants completed purchasing trials in an experimental marketplace, a virtual store designed to mimic real-world shopping environments. In each lab session, participants completed multiple trials in which the price of their assigned cigarette increased progressively from $0.13 in the first trial to $4.00 in the final trial, while prices for other products (e-cigarettes, e-liquid, nicotine gum, snus, lozenges, and dip) remained constant. The mean and standard deviation of quantity purchased in each trial were calculated for all prices and sessions 1, 2, and 3.
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 104.22 (89.69) | 29.64 (42.16)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 52.38 (53.34) | 47.41 (47.85)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 22.22 (26.45) | 61.77 (54.45)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 10.68 (14.35) | 68.58 (58.21)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 4.97 (7.08) | 78.83 (65.29)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 1.75 (2.90) | 79.02 (64.63)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 104.55 (70.02) | 28.32 (54.07)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 54.65 (56.45) | 39.37 (60.72)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 15.61 (25.92) | 89.70 (74.59)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 4.52 (9.06) | 94.11 (73.46)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 2.18 (4.61) | 97.91 (70.87)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 1.03 (2.60) | 98.73 (70.93)
  S3: Price $0.13 | 102.18 (90.28) | 21.36 (53.31)
  S3: Price $0.25 | 59.59 (57.12) | 38.84 (62.49)
  S3: Price $0.50 | 14.79 (22.88) | 80.79 (72.76)
  S3: Price $1.00 | 5.38 (9.75) | 83.03 (70.57)
  S3: Price $2.00 | 2.95 (5.91) | 93.66 (73.98)
  S3: Price $4.00 | 1.50 (2.88) | 87.03 (67.09)

2. Primary Outcome: Low Ventilated Cigarette Purchases
Description: Participants completed purchasing trials in an experimental marketplace, a virtual store designed to mimic real-world shopping environments. In each lab session, participants completed multiple trials in which the price of High Ventilated Cigarettes (HVC) increased progressively from $0.13 in the first trial to $4.00 in the final trial foe ventilated cigarette users and Low Ventilated Cigarettes (LVC) increased progressively from $0.13 in the first trial to $4.00 for the unventilated group, while prices for other products (Low Ventilated Cigarettes (LVC), e-cigarettes, e-liquid, nicotine gum, snus, lozenges, and dip) remained constant. The mean and standard deviation of quantity purchased in each trial was calculated for all prices and sessions 1, 2, and 3.
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 40.84 (58.73) | 123.91 (96.10)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 53.52 (64.66) | 70.39 (64.85)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 56.29 (62.22) | 28.89 (34.04)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 56.86 (66.67) | 9.36 (17.44)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 58.45 (63.78) | 3.33 (7.38)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 62.91 (61.87) | 0.97 (3.28)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 25.27 (44.72) | 127.92 (106.05)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 46.16 (56.88) | 77.08 (74.06)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 70.81 (62.72) | 13.86 (25.67)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 77.59 (61.05) | 5.21 (13.95)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 77.25 (60.82) | 1.73 (5.79)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 82.09 (61.17) | 0.76 (2.73)
  S3: Price $0.13 | 26.47 (56.64) | 122.76 (99.18)
  S3: Price $0.25 | 38.63 (58.61) | 60.65 (71.91)
  S3: Price $0.50 | 66.32 (62.23) | 8.97 (22.86)
  S3: Price $1.00 | 69.02 (61.75) | 1.94 (7.12)
  S3: Price $2.00 | 69.91 (61.74) | 0.32 (1.25)
  S3: Price $4.00 | 71.64 (60.94) | 0.11 (0.51)

3. Primary Outcome: E-Cigarette Purchases
Description: Participants completed purchasing trials in an experimental marketplace, a virtual store designed to mimic real-world shopping environments. In each lab session, participants completed multiple trials in which the price of High Ventilated Cigarettes (HVC) increased progressively from $0.13 in the first trial to $4.00 in the final trial for ventilated cigarette users and Low Ventilated Cigarettes (LVC) increased progressively from $0.13 in the first trial to $4.00 for the unventilated group, while prices for other products (Low Ventilated Cigarettes (LVC), e-cigarettes, e-liquid, nicotine gum, snus, lozenges, and dip) remained constant. The mean and standard deviation of quantity purchased in each trial was calculated for all prices and sessions 1, 2, and 3.
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 0.32 (0.70) | 0.47 (0.73)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 0.32 (0.67) | 0.44 (0.69)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 0.27 (0.65) | 0.52 (0.77)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 0.50 (1.13) | 0.86 (2.05)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 0.50 (1.02) | 0.91 (2.40)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 0.72 (1.32) | 1.16 (2.51)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 0.15 (0.56) | 0.27 (0.56)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 0.09 (0.47) | 0.22 (0.42)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 0.11 (0.49) | 0.27 (0.45)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 0.18 (0.65) | 0.29 (0.57)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 0.13 (0.63) | 0.29 (0.61)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 0.13 (0.63) | 0.29 (0.61)
  S3: Price $0.13 | 0.14 (0.51) | 0.08 (0.27)
  S3: Price $0.25 | 0.09 (0.47) | 0.16 (0.44)
  S3: Price $0.50 | 0.11 (0.62) | 0.24 (0.43)
  S3: Price $1.00 | 0.13 (0.63) | 0.29 (0.61)
  S3: Price $2.00 | 0.13 (0.63) | 0.29 (0.52)
  S3: Price $4.00 | 0.13 (0.63) | 0.32 (0.57)

4. Primary Outcome: E-liquid Purchases
Description: as for outcome 2
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 0.18 (0.81) | 0.31 (1.19)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 0.09 (0.36) | 0.08 (0.50)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 0.05 (0.21) | 0.13 (0.83)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 0.09 (0.36) | 0.19 (1.16)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 0.05 (0.21) | 0.25 (1.50)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 0.09 (0.36) | 0.22 (1.17)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 0.07 (0.45) | 0.08 (0.36)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 0.07 (0.45) | 0.08 (0.36)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 0.07 (0.45) | 0.08 (0.36)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 0.18 (0.87) | 0.08 (0.36)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 0.07 (0.45) | 0.13 (0.48)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 0.07 (0.45) | 0.11 (0.45)
  S3: Price $0.13 | 0.07 (0.45) | 0.21 (0.74)
  S3: Price $0.25 | 0.09 (0.60) | 0.15 (0.49)
  S3: Price $0.50 | 0.14 (0.90) | 0.10 (0.38)
  S3: Price $1.00 | 0.18 (1.21) | 0.10 (0.38)
  S3: Price $2.00 | 0.16 (1.05) | 0.10 (0.38)
  S3: Price $4.00 | 0.14 (0.90) | 0.10 (0.38)

5. Primary Outcome: Gum Purchases
Description: as for outcome 2
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 0.27 (0.89) | 0.39 (1.17)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 0.29 (0.90) | 0.17 (0.61)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 0.25 (0.97) | 0.25 (1.05)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 0.14 (0.41) | 0.39 (1.27)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 0.11 (0.39) | 0.39 (1.36)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 0.34 (1.23) | 0.31 (1.19)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 0.09 (0.60) | 0.08 (0.36)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 0.09 (0.60) | 0.03 (0.16)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 0.09 (0.60) | 0.0 (0.0)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 0.09 (0.60) | 0.37 (1.53)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 0.09 (0.60) | 0.05 (0.33)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 0.09 (0.60) | 0.73 (3.45)
  S3: Price $0.13 | 0.05 (0.30) | 0.00 (0.00)
  S3: Price $0.25 | 0.05 (0.30) | 0.00 (0.00)
  S3: Price $0.50 | 0.05 (0.30) | 0.26 (1.62)
  S3: Price $1.00 | 0.05 (0.30) | 0.00 (0.00)
  S3: Price $2.00 | 0.05 (0.30) | 0.05 (0.32)
  S3: Price $4.00 | 0.05 (0.30) | 0.32 (1.64)

6. Primary Outcome: Snus Purchases
Description: as for outcome 2
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 0.27 (1.81) | 0.33 (2.00)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 0.05 (0.30) | 0.28 (1.67)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 0.00 (0.00) | 0.00 (0.00)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 0.05 (0.30) | 0.11 (0.67)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 0.05 (0.30) | 0.00 (0.00)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 0.23 (0.15) | 0.17 (1.00)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 0.00 (0.00) | 0.27 (1.64)
  S3: Price $0.13 | 0.00 (0.00) | 1.31 (8.11)
  S3: Price $0.25 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $0.50 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $1.00 | 0.00 (0.00) | 1.31 (8.11)
  S3: Price $2.00 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $4.00 | 0.00 (0.00) | 1.36 (8.12)

7. Primary Outcome: Lozenge Purchases
Description: as for outcome 2
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 0.91 (4.34) | 0.31 (1.32)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 0.45 (3.02) | 0.22 (0.93)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 1.25 (6.01) | 0.11 (0.67)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 0.45 (3.02) | 0.19 (0.82)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 0.47 (3.02) | 0.28 (1.19)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 0.45 (3.02) | 0.22 (0.93)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 0.00 (0.00) | 0.00 (0.00)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $0.13 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $0.25 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $0.50 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $1.00 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $2.00 | 0.00 (0.00) | 0.00 (0.00)
  S3: Price $4.00 | 0.00 (0.00) | 0.00 (0.00)

8. Primary Outcome: Dip Purchases
Description: as for outcome 2
Time Frame: Week 2 (Session 1), Week 6 (Sessions 2), Week 10 (Session 3)
Population: There are a few data points missing for a couple of participants; therefore, the sample size may be slightly different.
Measure: Mean (Standard Deviation); unit: single unit quantity purchased
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
Number analyzed (Participants) | 44 | 38
single unit quantity purchased
  S1: Price $0.13: number analyzed (Participants) | 44 | 36
  S1: Price $0.13 | 0.07 (0.45) | 0.17 (1.00)
  S1: Price $0.25: number analyzed (Participants) | 44 | 36
  S1: Price $0.25 | 0.00 (0.00) | 0.00 (0.00)
  S1: Price $0.50: number analyzed (Participants) | 44 | 36
  S1: Price $0.50 | 0.14 (0.90) | 0.00 (0.00)
  S1: Price $1.00: number analyzed (Participants) | 44 | 36
  S1: Price $1.00 | 0.07 (0.33) | 0.06 (0.33)
  S1: Price $2.00: number analyzed (Participants) | 44 | 36
  S1: Price $2.00 | 0.05 (0.30) | 0.00 (0.00)
  S1: Price $4.00: number analyzed (Participants) | 44 | 36
  S1: Price $4.00 | 0.09 (0.60) | 0.00 (0.00)
  S2: Price $0.13: number analyzed (Participants) | 44 | 37
  S2: Price $0.13 | 0.00 (0.00) | 0.32 (1.97)
  S2: Price $0.25: number analyzed (Participants) | 44 | 37
  S2: Price $0.25 | 0.00 (0.00) | 0.22 (1.32)
  S2: Price $0.50: number analyzed (Participants) | 44 | 37
  S2: Price $0.50 | 0.00 (0.00) | 0.27 (1.64)
  S2: Price $1.00: number analyzed (Participants) | 44 | 37
  S2: Price $1.00 | 0.00 (0.00) | 0.05 (0.33)
  S2: Price $2.00: number analyzed (Participants) | 44 | 37
  S2: Price $2.00 | 0.00 (0.00) | 0.27 (1.64)
  S2: Price $4.00: number analyzed (Participants) | 44 | 37
  S2: Price $4.00 | 0.00 (0.00) | 0.49 (2.37)
  S3: Price $0.13 | 0.00 (0.00) | 0.39 (2.43)
  S3: Price $0.25 | 0.00 (0.00) | 0.55 (3.41)
  S3: Price $0.50 | 0.00 (0.00) | 0.55 (3.41)
  S3: Price $1.00 | 0.00 (0.00) | 0.61 (3.73)
  S3: Price $2.00 | 0.00 (0.00) | 0.66 (4.06)
  S3: Price $4.00 | 0.00 (0.00) | 0.68 (4.06)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Thank you for the clarification. Consistent with our previous ETM studies, Adverse Events are reported by study arm, not by individual product (e.g., Ventilated Cigarettes, Unventilated Cigarettes, E-cigarettes, Chew, etc.). All deaths, Serious Adverse Events, and Other Adverse Events meeting the reporting definitions are included in the Adverse Events module by arm accordingly. The interventions are the ventilation vs unventilated cigarettes.
Arm/Group | Ventilated Cigarettes | Unventilated Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/38
Other Adverse Events (participants affected / at risk) | 0/44 | 0/38

LIMITATIONS AND CAVEATS:
During the study, the researchers detected changes in the ventilation levels of the low-ventilated study cigarettes introduced by the manufacturer, which may have altered the intended intervention and results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT03306173/Prot_003.pdf
  • Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03306173/SAP_004.pdf